CLINICAL TRIAL: NCT02336386
Title: Study of Cyclophosphamide，Liposome Doxorubicin Dexamethasone（CDD) Plus Bortezomib Compared With CDD in the Relapsed or Refractory Multiple Myeloma Combined With Extramedullary Plasmacytoma Patients
Brief Title: CDD Plus Bortezomib or CDDin Relapsed or Refractory Multiple Myeloma With Extramedullary Plasmacytoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yuping Zhong, Chief physician, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMA-MM
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Extramedullary Plasmacytoma
Keywords: Bortezomib
MeSH Terms: interventions — Cyclophosphamide; Dexamethasone; Bortezomib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CDD Plus Bortezomib (Experimental): Patients will receive Bortezomib (1.3mg/m2) Subcutaneous injection on Days 1, 4,8,11 and plus dexamethasone 20 mg/day PO on Days 1-4, 9-12,Cyclophosphamide 300mg/m2 D1-4, Liposome doxorubicin 40mg D4 of each 28-day cycle; Patients may continue to receive treatment until PD or unacceptable toxicity.
  Interventions: Drug: CDD Plus Bortezomib
- CDD (Active Comparator): Dexamethasone 20 mg/day PO on Days 1-4, 9-12,Cyclophosphamide 300mg/m2 D1-4, doxorubicin Dexamethasone 40mg D4 of each 28-day cycle; Patients may continue to receive treatment until PD or unacceptable toxicity
  Interventions: Drug: CDD

INTERVENTIONS:
Drug: CDD — Chemotherapy
  Other Names: Cyclophosphamide,Liposome doxorubicin and Dexamethasone
  Arms: CDD
Drug: CDD Plus Bortezomib — Chemotherapy plus Proteasome Inhibitors
  Other Names: Chemotherapy Plus Bortezomib
  Arms: CDD Plus Bortezomib

SUMMARY:
The purpose of this study is to determine whether Cyclophosphamide, Liposome doxorubicin and Dexamethasone（CDD) Plus Bortezomib might have effective in extramedullary plasmacytoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients from 18 to 80
* Biopsy-proven EMP with relapsed or refractory Myeloma disease. Patients may be proteasome inhibitor-exposed or naive, but cannot be refractory to proteasome inhibitor therapy
* Disease requiring further treatment
* Measurable disease such as M protein and Objective and measurable of EMP
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2
* Meet the clinical laboratories criteria as specified in the protocol
* Voluntary written consent

Exclusion Criteria:

* Female patients who are lactating, breastfeeding or pregnant
* Evidence of current uncontrolled cardiovascular conditions as specified in study protocol
* Requirement for other concomitant chemotherapy, immunotherapy, radiotherapy, which would be considered as a treatment of EMP.
* Comorbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Ongoing or active infection, known HIV positive, active hepatitis B or C infection
* Psychiatric illness/social situations that would limit compliance with study requirements
* Known allergy to any of the study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with overall hematologic response | Assessed every 2 cycles (median length of the endpoint assessment period is projected to be approximately 24 months)
  Complete response, very good partial response and partial response

SECONDARY OUTCOMES:
Number of patients with EMP response | Assessed every 2 cyeles period is projected to be approximately 24 months
  response rate
Overall survival | Monthly up to 3 years
  The median overall survival
Time from diagnosis ofEMP to the date of death | Monthly up to 3 years
Progression free survival | Monthly up to 2 years
Time from date of diagnosis of EMP to the date of first documentation of disease | Monthly up to 2 years
Number of adverse events | Monthly up to 3 years
  Adverse events, serious adverse events, assessment of clinical laboratory values from the date of signing of the informed consent form through 30 days after the last dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Yuping Zhong, Doctor, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Yuping ZHONG, Beijing, Beijing Municipality, China